CLINICAL TRIAL: NCT02287948
Title: Validation Study for Using Wii FIT Balance Board to Recording Balance Parameters in Healthy Subjects and Multiple Sclerosis Subjects
Brief Title: Wii FIT Balance Board to Recording Balance Parameters in Multiple Sclerosis Subjects
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, MD, University Hospital of Ferrara
Other Study IDs: WII Balance Board_MS
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Postural Balance; Multiple Sclerosis
Keywords: Balance; Multiple Sclerosis; Nintendo Wii Fit
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MS subjects group: Multiple sclerosis subjects wiht mild-moderate gait disability with EDSS score not higher than 5.5
  Interventions: Device: Nintendo Wii Fit Balance Board
- Healthy subjects group: Healthy subjects age-matched with multiple sclerosis subjects.
  Interventions: Device: Nintendo Wii Fit Balance Board

INTERVENTIONS:
Device: Nintendo Wii Fit Balance Board — Clinical and instrumental evaluations carry out on the same day.
  1) Instrumental evaluations
  All subjects (healthy + MS) will ask to perform the following tasks both on force platform and Wii Fit Balance Board:
  * Open eyes, monopodalic balance for 20 seconds
  * Closed eyes, monopodalic balance for 20 seconds
  * Open eyes, balance on both feet for 60 seconds
  * Closed eyes, balance on both feet for 60 seconds
  During trials subjects can leave arms in the most comfortable position they prefere
  Subjects will perform every task for 5 times; they can rest for 30 seconds between every trials.

SUMMARY:
Balance disorders are frequently observed in patients with Multiple Sclerosis (MS) and the deterioration of the static and dynamic control of balance is an important and basic symptom of disease progression.

Measure balance disorders with force platforme requires personnel and represent a significant cost.

The platform Nintendo Wii Fit represents a valid economic alternative

DETAILED DESCRIPTION:
Balance disorders are frequently observed in patients with MS and are the most disabling symptoms; in subjects with moderate disabilities for balance, the deterioration of the static and dynamic control of balance is an important and basic symptom of disease progression.

From a clinical point of view, the reliability of being able to discriminate patients who have the highest probability of falling than those with lower probability is crucial to develop a program aimed at the prevention of falls.

Potentially the parameters measured wiht torque platform can be an objective, reliable and accurate for discriminating patients with the highest probability of falling than those with low probability, and may be useful to highlight the deficits and improvements in the ability to maintain balance after specific rehabilitation. However posturographic systems represent a significant cost, require a dedicated and qualified personnel to use. A possible solution to not use force platforms could be the implementation of software to interface with the Nintendo Wii Fit Balance Board (WBB) with a personal computer.

The platform Nintendo Wii Fit presents a set of sensors lower compared to a traditional force platform, but can represent a valid economic alternative to more complex systems, in addition to being already used as a rehabilitation tool in the literature in more than one study. Studies in healthy subjects have valid information on the study of the center of pressure (COP) obtained from WBB showing that the path lengths of the COP obtained from the WBB were valid and well correlated with those recorded by a dynamometric platform.

ELIGIBILITY:
Inclusion Criteria (Healthy subjects):

* Male and female, aged > 18, < 80 years;
* healthy.

Exclusion Criteria (Healthy subjects):

* pregnancy;
* previous diagnosis of debilitating diseases;
* previous diagnosis of orthopedic, neurological, vestibular or that may affect the balance.

Inclusion Criteria (Multiple Sclerosis subjects):

* Male and female, aged > 18, < 80 years;
* subjects with a diagnosis of MS according to the McDonald criteria in course with relapse and remission, progressive, primary or secondary are included in the study;
* absence of disease exacerbations in the 3 months prior to enrollment;
* mild or moderate gait disability identified with the Expanded Disability Status Scale (EDSS) score not higher than 5.5. This degree of severity refers to a subject with restriction ambulatory activity but which does not require constantly an unilateral support (stick, crutch, other) for walking.

Exclusion Criteria (Multiple Sclerosis subjects):

* cognitive impairment assessed with Mini Mental Status Examination (MMSE) <24;
* neurological diseases associated with MS with possible involvement of motor functions;
* of internal conditions that might interfere with the ability to complete the study protocol in a secure manner;
* severe cognitive-behavioral (score less than 24 on the Mini Mental Status Examination);
* pregnancy;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Will be recruited 20 healthy subjects and 20 subject with a diagnosis of multiple sclerosis and mild to moderate disability ambulatory identified with a value not higher than 5.5 EDSS score. The subjects of both groups will be age-matched to exclude differences caused by age posturographic. All individuals carry out the task of torque balance both on the platform and on the Wii Fit Balance Board on the same day.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Parameters related with postural balance and the chance to fall | one evaluation in one day
  Instrumental evaluations carry out on the same day.
  All subjects will perform the following tasks both on force platform and Wii Fit Balance Board:
  * Open eyes, monopodalic balance for 20 seconds
  * Closed eyes, monopodalic balance for 20 seconds
  * Open eyes, balance on both feet for 60 seconds
  * Closed eyes, balance on both feet for 60 seconds
  During trials subjects can leave arms in the most comfortable position they prefere Subjects will perform every task for 5 times; they can rest for 30 seconds between every trials.

SECONDARY OUTCOMES:
Timed "up and go" test (TUG) | one evaluation in one day
  Timed "up and go" test validity has been demonstrated with Berg Balance test correlation, gait speed and ability to step on the stairs; this test has been recently validated for multiple sclerosis subjects evaluation.
Dynamic Gait Index (DGI) | one evaluation in one day
  DGI indicates the subject's ability to adapt walking patterns according to environmental changes (ie changes in the speed, turn the head, climb over or around obstacles or stairs). The DGI was created to assess the balance dysfunction in individuals with alterations in the way of vestibular apparatus, but it represents a reliable assessment scale for subjects with multiple sclerosis (McConvey 2005).
Berg Balance Scale | one evaluation in one day
  This scale tests static and dynamic activities. The level of each item has a score range 0-4 determined the ability of the patient to the ability to perform the task tested. The results of each item are added together, the total score is 56.
Unified Balance Scale - Unified Balance Scale (UBS) | one evaluation in one day
  The 27 items that make up the UBS are part of the existing three scales: Berg Balance Sclale (BBS), Performance Oriented Mobility Scale (Scale and Tinetti POMA) and Fullerton Advanced Balance Scale (FABS).

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, Principal Investigator — Ospedale San Giorgio
Locations (1):
- Ferrara University Hospital, Ferrara, Ferrara, Italy